CLINICAL TRIAL: NCT03857581
Title: Clozapine Versus Olanzapine as Treatment for Comorbid Psychotic Disorder and Substance Use Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Sandarsh Surya, Assistant Professor, Department of Psychiatry and Health Behavior, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1303985
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Psychosis; Substance Use Disorders
Keywords: Schizophrenia; Schizoaffective disorder; Bipolar disorder; Major depressive disorder; Psychosis; Substance abuse; Clozapine; Olanzapine
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major | interventions — Clozapine; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clozapine Arm (Experimental)
  Interventions: Drug: Clozapine
- Olanzapine Arm (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Clozapine — Subjects will be randomly assigned to clozapine or olanzapine and followed for up to 12 weeks with weekly visits.
  Arms: Clozapine Arm
Drug: Olanzapine — Subjects will be randomly assigned to clozapine or olanzapine and followed for up to 12 weeks with weekly visits.
  Arms: Olanzapine Arm

SUMMARY:
The purpose of this trial is to determine if patients with comorbid psychotic disorder and substance use disorder will continue in treatment longer if treated with clozapine than with olanzapine, and will have greater reductions in psychosis and in substance use if treated with clozapine than treated with olanzapine. The specific aims and hypotheses of this trial are: 1. To compare the enduring effectiveness and tolerability of clozapine and olanzapine, as measured by time to all-cause treatment discontinuation, over 12 weeks of follow-up; The investigators hypothesize that patients assigned to clozapine treatment will have significantly longer times to all cause treatment discontinuation, 2. To compare the total psychosis items scores between patients treated with clozapine and patients treated with olanzapine over 12 weeks of follow-up; The investigators hypothesize that patients treated with clozapine will have significantly lower total psychosis items scores than patients treated with olanzapine, and 3. To compare the frequencies of positive urine drug screens and blood alcohol levels (obtained weekly throughout 12 weeks of follow-up) between patients treated with clozapine and patients treated with olanzapine; The investigators hypothesize that patients treated with clozapine will have significantly fewer positive urine drug screens and blood alcohol levels than patients treated with olanzapine.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age, male or female (post-menopausal, surgically sterilized, or receiving either one of the listed contraception - depot contraceptive, Intrauterine device, or implanted hormonal contraceptive),
* who meet DSM-V criteria for schizophrenia, schizoaffective disorder, bipolar disorder with psychotic features, depression with psychotic features, or delusional disorder, and have ratings of Moderate or greater on at least one of the Brief Psychiatric Rating Scale psychosis items,
* who meet DSM-V criteria for at least one of alcohol, marijuana, cocaine, stimulant, or opioid use disorder, and have an admission urine drug screen positive for at least one of these substances,
* who have a stable living situation (family or supervised living, e.g. personal care home) to return to after release into the community,
* and who provide signed informed consent to participate (after testing for comprehension).

Exclusion Criteria:

* Prior failure to respond or tolerate clozapine or olanzapine
* Logistics that prevent outpatient follow-up at Serenity Behavioral Health Adult Outpatient services

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Frequencies of positive urine drug screens and breathalyzer alcohol levels | 12 weeks
  Participants will have weekly urine drug screens and alcohol level measurement using breathalyzer to monitor ongoing substance and alcohol abuse.

SECONDARY OUTCOMES:
All-cause treatment discontinuation | 12 weeks
  Discontinuation rate due to any cause (treatment non-compliance, worsening of mental health conditions, withdrawal of consent)
Brief Psychiatric Rating Scale (BPRS) - Positive Psychopathology items | 12 weeks
  BPRS scale is used to measure and monitor for symptoms of schizophrenia. For the purpose of the study, we will be measuring 4 items to monitor for positive psychopathology. The items are
  1. Suspiciousness
  2. Hallucinations
  3. Unusual thought content
  4. Conceptual disorganization
  Each item is rated on a scale of 1 to 7. 1 being condition not present and 7 being extreme form of the condition present. The maximum score a participant can score is 28 and minimum score is 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Sandarsh Surya, Evans, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided